CLINICAL TRIAL: NCT03076762
Title: Comparative Study of the Efficacy and Safety Between Suburothelial and Trigonal Intravesical Botulinum Toxin A Injection in Treatment of Interstitial Cystitis Refractory to Conventional Treatment - A Prospective, Randomized, Clinical Trial
Brief Title: Comparative Study Suburothelial and Trigonal Botulinum Toxin A Injection in Treatment of Interstitial Cystitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Chairman, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BuddhistTCGH2003-01
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Bladder Pain Syndrome
Keywords: interstitial cystitis; pain; intravesical injection; therapy; bladder
MeSH Terms: conditions — Cystitis, Interstitial; Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to receive intravesical injection of 100U of BoNT-A (BOTOX, Allergan, Irvine, CA, USA) into the trigone (the treatment group) or suburothelium (the comparative group) immediately followed by cystoscopic hydrodistention under intravenous general anesthesia in the operation room.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigator and outcome assessor are blinded to the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravesical suburothelial injection (Experimental): Patients assigned for suburothelial injections received 100 U of onabotulinumtoxinA in 20 sites injected in the bladder body on treatment day and follow-up
  Interventions: Drug: intravesical onabotulinumtoxinA injection
- Intravesical trigonal injection (Active Comparator): Patients assigned trigonal injections will receive 100U of onabotulinumtoxinA at 10 sites injected at the trigonal area (5 injections behind interureteric ridge and 5 inside the trigone) on treatment day and follow-up.
  Interventions: Drug: intravesical onabotulinumtoxinA injection

INTERVENTIONS:
Drug: intravesical onabotulinumtoxinA injection — Each vial of onabotulinumtoxinA will be diluted with 10 ml of normal saline, resulting in 10U onabotulinumtoxinA per 1.0 ml. Patients assigned for suburothelial BoNT-A injections received 20 injections in the bladder body whereas those assigned trigonal injections will receive 10 sites injections at the trigonal area (5 injections behind interureteric ridge and 5 inside the trigone).
  Other Names: BOTOX

SUMMARY:
There is no consensus of the therapeutic efficacy and safety between suburothelial injection and trigonal injection of botulinum toxin A (BoNT-A) in treatment of interstitial cystitis/bladder pain syndrome (IC/BPS) It is unmet to clarify which injection method is superior in clinical efficacy and patient safety. This study was designed in a randomized, double-blind trial to test the therapeutic effects and adverse events between intravesical BoNTA injection into suburothelium and trigone. The results of this study might provide clinical evidence for a better therapeutic regimen of BoNT-A in the treatment of IC/PBS.

DETAILED DESCRIPTION:
Introduction Interstitial cystitis/painful bladder syndrome (IC/PBS) is a debilitating chronic disease of unknown etiology characterized by urgency frequency and suprapubic pain at full bladder. Current treatments are usually unsuccessful in completely eradicating bladder pain and increasing bladder capacity. Intravesical resiniferatoxin once was considered to be effective but this has not been shown in a large scale multiple center trial. Several oral medication such as pentosanpolysulphate (PPS), amitryptynine, cyclosporin have been tried but the therapeutic efficacy have been proven ineffective. Intravesical treatment with heparin, hyaluronic acid, chondroitin sulphate, bacillus Calmette-Guerin, dimethylsulphoxide, resiniferatoxin, or botulinum toxin A has been shown early effectiveness in some patients. However, the placebo effect should be weighed and randomized, double-blind trials should be undertaken to demonstrate the actual therapeutic effects of these therapeutic modalities.

Although botulinum toxin type A (BoNT-A) has been widely reported in its efficacy in the treatment of neurogenic and idiopathic detrusor overactivity (DO) with satisfactory results, there have only been few studies using BoNT-A in treatment of IC/PBS. In recent basic researches, BoNT-A has been shown to inhibit not only the release of acetylcholine and norepinephrine, but also that of nerve growth factor, adenosine triphosphate, substance P and calcitonin gene-related peptide from the nerve fibers and urothelium. In clinical experiments, BoNT-A has been shown to reduce DO, impaired bladder sensation, and decrease visceral pain in chronic inflammatory diseases. These results suggest that BoNT-A treatment can modulate sensory transmission as well as reduce detrusor contractility. Although BoNT-A injection seems promising in treating symptoms of IC/PBS, long term results did not provide successful outcome. The limited successful result is possibly due to inadequate distribution of BoNT-A delivered to the bladder wall, inadequate dose of toxin, or lacking of some promoting factors to enhance the therapeutic effect of BoNT-A. Repeated intravesical BoNT-A injections was recently performed in refractory IC/PBS and the therapeutic effects seems promising. About 70% of the patients with non-ulcer type IC/PBS may benefit from repeated BoNT-A injections every 6 months. Immunohistochemistry study also confirmed the reduction of inflammatory biomarkers and pro-apoptotic proteins such as Bax and Bad expressions after repeated BoNT-A injections.

Concerning the injection sites of BoNT-A for IC/BPS bladders, there is no consensus. Suburothelial injection and Trigonal injection have all been used in treatment of IC/BPS and the short-term and long-term results are equivalent. It is unmet to clarify which injection method is superior in clinical efficacy and patient safety. This study was designed in a randomized, double-blind trial to test the therapeutic effects and adverse events between intravesical BoNTA injection into suburothelium and trigone. The results of this study might provide clinical evidence for a better therapeutic regimen of BoNT-A in the treatment of IC/PBS.

Materials and Methods

A total of 60 patients with IC/PBS who have failed previous treatments for at least 6 months will be enrolled in this study. A diagnosis of IC/PBS has been established based on characteristic symptoms and cystoscopic findings of glomerulations, petechia, or mucosal fissures after hydrodistention. All patients have been treated with at least two types of treatment modalities including non-steroid anti-inflammatory drugs, oral PPS, intravesical instillation of heparin, hyaluronic acid, or tricyclic antidepressant for at least 6 months but the symptoms remained unchanged or relapsed. They will be investigated thoroughly on enrollment and will be excluded if not meeting the inclusion criteria of NIDDK. However, in this study the patients with Hunner's ulcer will not be included because previous study has shown that ulcer type IC/BPS does not respond to intravesical BoNT-A injection.

Patients will be requested to keep a 3-day voiding diary prior to treatment to record the functional bladder capacity (FBC) and the number of urinary frequency and nocturnal. The IC symptoms will be assessed by the O'Leary-Sant symptom and problem indexes. The pain score will be reported by patient self-assessment using a 10-point visual analog scale (VAS) system. Videourodynamic study and potassium chloride (KCl) sensitivity test will be routinely performed and patients will be informed of the possible complications associated with BoNT-A injection such as generalized muscle weakness, difficult urination, transient urinary retention, or urinary tract infections.

Videourodynamic study will be performed by standard procedures using a 6 Fr dual channel catheter and an 8 Fr rectal balloon catheter. Cystometric study will be performed with normal saline at a filling rate of 20 ml/min. All descriptions and terminology in this report are in accordance with the recommendations of the International Continence Society. After the videourodynamic study, 40ml KCl solution of 0.4M will be infused slowly into the bladder and the test will be regarded as positive when painful (of ≧2 VAS score) or urgency sensation (urgency severity score increased by ≧1) is elicited compared to normal saline infusion during urodynamic study.

This study will be performed in Hualien Tzu chi General.The study should be approved by the Institutional Review Board (IRB) and ethics committee of the university and will be registered in ClinicalTrial.gov. Each patient will be informed about the study rationale and procedures, and written, informed consent will be obtained before treatment.

Eligible patients will be admitted for the treatment. They will be randomly assigned to receive intravesical injection of 100U of BoNT-A (BOTOX, Allergan, Irvine, CA, USA) into the trigone (the treatment group) or suburothelium (the comparative group) immediately followed by cystoscopic hydrodistention under intravenous general anesthesia in the operation room. Blood (10ml) and urine samples (30ml) will be collected before intravesical injection and after bladder hydrodistention. Bladder wall biopsies will also be performed after hydrodistention. The patients will be allocated to treatment or control group by the permuted block randomization code which is centrally controlled by a clinical pharmacist who prepares the solution for injection. The intravesical injection was performed by a urology attending doctor without recording the injection mode in the medical chart. The principle investigator, patients, and study nurse did not know the injection mode to the patients' bladder to keep the study in a double-blind condition.

Each vial of BoNT-A will be diluted with 10 ml of normal saline, resulting in 10U BoNT-A per 1.0 ml. Patients assigned for suburothelial BoNT-A injections received 20 injections in the bladder body whereas those assigned trigonal injections will receive 10 sites injections at the trigonal area (5 injections behind interureteric ridge and 5 inside the trigone). The injection needle will be inserted about 1mm into the urothelium at the bladder wall, using a 23 gauge needle and rigid cystoscopic injection instrument (22 Fr, Richard Wolf, and Knittlingen, Germany). Cystoscopic hydrodistention will be performed to an intravesical pressure of 80 cm water for 15 minutes and the maximal bladder capacity (MBC) under hydrodistention will be recorded. Bladder biopsies will be taken at the four sites about 2cm lateral and posterior to the ureteral orifice after hydrodistention.

After the BoNT-A injections, a 14 Fr urethral Foley catheter will be indwelled for one night and patients will be discharged on the next day. Oral antibiotics will be prescribed for 7 days. Patients will be followed up in the outpatient clinic 2 weeks and 4 weeks later. Then the patients will be followed up at out-patient clinic at 2 weeks, 4 weeks and 8 weeks.

Data from the 3-day voiding diary and symptom inventory using the O'Leary-Sant symptom score, as well as information on FBC, daily urinary frequency, nocturia, and pain VAS will be recorded at baseline, 2 weeks, 4 weeks, and 8 weeks. The largest voided volume in the 3-day voiding diary will be considered as a measure of FBC. At 8-week follow-up after the intravesical injection patients will be questioned of the current bladder condition and a urodynamics study with KCl test will be performed.

The urodynamic study will be performed at baseline and 12 weeks after intravesical treatment. The urodynamic parameters include first sensation of bladder filling (FSF), urge sensation (US), cystometric bladder capacity (CBC), detrusor pressure (Pdet), maximum flow rate (Qmax) during voiding and postvoid residual (PVR). KCl test will also be performed.

The primary end-point of this study is the reduction of bladder pain at 8-week follow-up. If patient has a reduction of VAS pain score of 2 or more, they will be considered as successfully treated. The treatment outcome will also be assessed by the global response assessment (GRA) to evaluate the overall perception of treatment result. The result will be considered as excellent when patients report improvement in the GRA by >2 or patients become free of bladder pain (VAS=0). The outcome will be considered improved if there is improvement in the GRA by =1. Patients with excellent and improved results will be considered as having subjectively successful result.

The results of voiding diary, urodynamic study, IC symptom score and pain VAS will be compared between baseline and 8-week end-point. Long-term successful results will be assessed by self-reported improved GRA and pain VAS at 6 months and further. Data will be compared between treatment and placebo groups. A p-value of less than 0.05 will be considered statistically significant.

If patients still feel bladder pain and unsuccessful results at the end-point, repeated BoNT-A injection will be given at 3 months in the same procedure. At the same time, bladder biopsy, urine and blood samples will also be collected for further study. . If patient does not want to receive repeat BoNT-A injection, intravesical hyaluronic acid instillations will be proceeded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have been diagnosed as IC/BPS based on characteristic symptoms and cystoscopic findings of glomerulations, petechia, or mucosal fissures after hydrodistention
2. Patients have been treated with at least two types of treatment modalities including non-steroid anti-inflammatory drugs, oral PPS, intravesical instillation of heparin, hyaluronic acid, or tricyclic antidepressant for at least 6 months but the symptoms remained unchanged or relapsed.
3. Patients who have bladder pain VAS of 3 or greater

Exclusion Criteria:

1. Patients conditions not meeting the inclusion criteria of NIDDK
2. Patients with Hunner's ulcer
3. Patients with active urinary tract infection
4. Patients who cannot keep a 3-day voiding diary prior to treatment
5. Patients who do not sign informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Reduction of bladder pain visual analog scale (VAS) | baseline to 8 weeks
  Evaluation of the change of VAS from baseline to 8 weeks

SECONDARY OUTCOMES:
Interstitial cystitis symptom index (ICSI) | baseline to 8 weeks
  Evaluation of the change of ICSI froim baseline to 8 weeks
Functional bladder capacity | baseline to 8 weeks
  The change of maximal bladder capacity in voiding diary from baseline to 8 weeks
Maximum flow rate (Qmax) | baseline to 8 weeks
  The change of Qmax from baseline to 8 weeks
Voided volume | baseline to 8 weeks
  Thde change of voided volume from baseline to 8 weeks
Postvoid residual volume | baseline to 8 weeks
  The change of postvoid residual volume from baseline to 8 weeks
Interstitial cystitis problem index (ICPI) | baseline to 8 weeks
  Evaluation of the change of ICPI from baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng HC Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital, Hualien
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Jiang YH, Jhang JF, Lee CL, Kuo HC. Comparative study of efficacy and safety between bladder body and trigonal intravesical onabotulinumtoxina injection in the treatment of interstitial cystitis refractory to conventional treatment-A prospective, randomized, clinical trial. Neurourol Urodyn. 2018 Apr;37(4):1467-1473. doi: 10.1002/nau.23475. Epub 2018 Jan 13. PMID 29331031